CLINICAL TRIAL: NCT01927120
Title: In Vivo Treg Expansion and Graft-Versus-Host Disease Prophylaxis With IL-2, Sirolimus, and Tacrolimus Following Allogeneic Hematopoietic Cell Transplantation
Brief Title: In Vivo Treg Expansion and Graft-Versus-Host Disease Prophylaxis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MCC-17578; NCI-2014-00755 (Other: NCI CTRP)
Record Dates: First submitted 2013-08-16; First posted 2013-08-22 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-03

CONDITIONS: Graft-Versus-Host-Disease
Keywords: GVHD; Allogeneic; Hematopoietic Cell Transplant
MeSH Terms: conditions — Graft vs Host Disease | interventions — Interleukin-2; aldesleukin; Tacrolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- GVHD Regimen (Experimental): Graft versus host disease (GVHD) prophylaxis regimen IL-2 with Sirolimus and Tacrolimus after allogeneic hematopoietic cell transplant (HCT).
  Interventions: Drug: IL-2; Drug: Tacrolimus; Drug: Sirolimus

INTERVENTIONS:
Drug: IL-2 — A subcutaneous injection will be administered 3 times a week (separated by at least 1 day between injections), from day 0 to +90 (+/- 7 days).
  Other Names: Proleukin®; (aldesleukin)
Drug: Tacrolimus — Will be administered at 0.01 mg/kg/day (based on ideal body weight) continuous IV infusion or equivalent oral dosing starting on day -3
Drug: Sirolimus — Orally on day -1. The dose for loading is 12 mg by mouth (PO)
  Other Names: Rapamune

SUMMARY:
IL-2 add-back post allogeneic hematopoietic stem cell transplant (HSCT), combined with Sirolimus (SIR), Tacrolimus (TAC) will optimize Treg reconstitution and prevent graft versus host disease (GVHD).

DETAILED DESCRIPTION:
1) Determine if a GVHD prophylaxis regimen of IL-2/SIR/TAC enhances in vivo Treg differentiation and growth; 2) Study the safety and effects of IL-2/SIR/TAC on the incidence of acute and chronic GVHD; 3) Evaluate the influence of dual IL-2 supplementation and mammalian target of rapamycin (mTOR) inhibition on T cell-specific signaling pathways and the polarization of emerging T helper cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have an available 8/8 human leukocyte antigen (HLA)-A, -B, -C, and -DRB1 matched-related or unrelated donor allogeneic hematopoietic peripheral blood stem cell graft.
* Acute myeloid leukemia, myelodysplasia, acute lymphoblastic leukemia, chronic myeloid leukemia, or myeloproliferative neoplasms requiring a matched allogeneic HSCT.

  * Acute Leukemia (AML or ALL) must be in complete remission defined as: <5% marrow blasts with no morphologic evidence of leukemia, no peripheral blasts, marrow >20% cellular, and peripheral absolute neutrophil count >1000/µL (platelet recovery is not required).
  * Myelodysplasia (MDS) and chronic myeloid leukemia (CML): Must have <5% marrow blasts.
  * Myeloproliferative neoplasms (MPN): Must have <5% peripheral / marrow blasts.
* Adequate vital organ function:

  1. Left ventricular ejection fraction (LVEF) ≥ 45% by multi gated acquisition (MUGA) scan or ECHO
  2. Forced expiratory volume at one second (FEV1), forced vital capacity (FVC), and adjusted diffusing lung capacity oxygenation (DLCO) ≥ 50% of predicted values on pulmonary function tests
  3. Transaminases (AST, ALT) < 2 times upper limit of normal values
  4. Creatinine clearance ≥ 50 cc/min.
* Performance status: Karnofsky Performance Status Score ≥ 80%
* Donor eligibility: Eligible donors will include healthy sibling, relative or unrelated donors that are matched with the patient at HLA-A, B, C, and DRB1 by high resolution typing.

Exclusion Criteria:

* Active infection not controlled with appropriate antimicrobial therapy
* History of HIV, hepatitis B, or hepatitis C infection
* Anti-thymocyte globulin, alemtuzumab, bortezomib, or cyclophosphamide administered within 14 days before or planned to receive with HCT conditioning or as part of GVHD prophylaxis in the 14 days after HCT.
* Hypersensitivity to recombinant human IL-2
* Chronic lymphocytic leukemia, Hodgkin lymphoma, and non-hodgkin lymphoma are excluded as these malignancies may express the IL-2 receptor and pose a potential growth signal to any present disease.
* Sorror's co-morbidity factors with total score >4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03-25 (Actual); Primary Completion 2016-08-25 (Actual); Study Completion 2017-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Betts, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Betts BC, Pidala J, Kim J, Mishra A, Nishihori T, Perez L, Ochoa-Bayona JL, Khimani F, Walton K, Bookout R, Nieder M, Khaira DK, Davila M, Alsina M, Field T, Ayala E, Locke FL, Riches M, Kharfan-Dabaja M, Fernandez H, Anasetti C. IL-2 promotes early Treg reconstitution after allogeneic hematopoietic cell transplantation. Haematologica. 2017 May;102(5):948-957. doi: 10.3324/haematol.2016.153072. Epub 2017 Jan 19. PMID 28104702
- See also: H. Lee Moffitt Cancer Center & Research Institute — http://www.moffitt.org
- See also: IL-2 promotes early Treg reconstitution after allogeneic hematopoietic cell transplantation — http://www.haematologica.org/content/early/2017/01/19/haematol.2016.153072.long

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Moffitt Cancer Center, April 2014 through December 2015.
Period: Overall Study
Arm/Group | GVHD Regimen
Started | 20
Completed | 10
Not Completed | 10

BASELINE CHARACTERISTICS:
Population: All participants.
Arm/Group | GVHD Regimen
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 49 [22 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Regulatory T Cells (Tregs)/Total CD4+ Cells at Day 30 Post-HCT
Description: Percentage of Treg among blood CD4+ T cells at day 30 after hematopoietic cell transplantation (HCT), to compare to SIR/TAC alone data from a previous trial (median of 16%). The study was designed to capture an increase in regulatory T cells from a median of 16.0% at day +30.
Time Frame: 30 days post HCT
Population: All participants.
Measure: Median (Full Range); unit: percentage of CD4+Tregs
Arm/Group | GVHD Regimen
Number analyzed (Participants) | 20
percentage of CD4+Tregs | 23.8 [12.8 to 39.3]

2. Secondary Outcome: Overall Survival at Day +365
Description: Overall survival will be defined as the time from transplant date to death from any cause.
Time Frame: 365 days post HCT
Population: All participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GVHD Regimen
Number analyzed (Participants) | 20
percentage of participants | 77.1 [49.3 to 90.7]

3. Secondary Outcome: Cumulative Incidence of Relapse
Description: Incidence of primary disease relapse per standard definitions.
Time Frame: 1 year post HCT
Population: All participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GVHD Regimen
Number analyzed (Participants) | 20
percentage of participants | 35.2 [9.2 to 63.3]

4. Secondary Outcome: Cumulative Incidence of Grade II-IV Acute GVHD by Day +100
Description: Acute GVHD will be graded per the 1995 consensus guidelines.
Time Frame: 100 days post HCT
Population: All participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GVHD Regimen
Number analyzed (Participants) | 20
percentage of participants | 40 [15.8 to 63.4]

5. Secondary Outcome: Cumulative Incidence of Chronic GVHD by Day +365
Description: Cumulative incidence of chronic GVHD by day +365 per NIH Consensus criteria.
Time Frame: 365 days post HCT
Population: All participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GVHD Regimen
Number analyzed (Participants) | 20
percentage of participants | 61.5 [36.1 to 79.3]

6. Secondary Outcome: Incidence of Non-relapse Death
Description: Incidence of Non-relapse death/Transplant-related mortality. Non-relapse death is defined as death in continuous remission from primary disease requiring transplantation.
Time Frame: 365 days post HCT
Population: All participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GVHD Regimen
Number analyzed (Participants) | 20
percentage of participants | 5.0 [0.0 to 65.6]

7. Secondary Outcome: Incidence of Unexpected or Serious Adverse Events (AEs)
Description: Grade 3-5 unexpected or serious adverse events (AEs) according to Common Terminology Criteria for Adverse Events (CTCAE) v.4.03) were captured up to day +130 or 30 days after the last dose of IL-2. Events listed, with causality in relation to study treatment noted.
Time Frame: Up to days 130 post HCT
Population: All participants.
Measure: Number; unit: adverse events
Arm/Group | GVHD Regimen
Number analyzed (Participants) | 20
adverse events
  VOD, possibly related | 2
  Portal vein thrombosis, possibly related | 1
  Sepsis, unlikely to be related | 1
  GI bleed, unrelated | 1
  Acute kidney injury, unrelated | 3
  Kidney stone, unrelated | 1
  Intracranial hemorrhage, unrelated | 1

8. Secondary Outcome: Proportion of Treg Among Blood CD4+ T Cells at Day +90 After HCT
Description: The proportion of Tregs to non-Treg CD4+ cells to be assessed at day +90. Natural Killer Cells (NKs): Median K/uL NK cells.
Time Frame: 90 days post HCT
Population: All participants.
Measure: Median (Full Range); unit: K/uL NK cells
Arm/Group | GVHD Regimen
Number analyzed (Participants) | 20
K/uL NK cells | 0.212 [0.079 to 0.605]

9. Secondary Outcome: STAT3, STAT5 (Y694), and S6 Phosphorylation Among Treg and Non-Treg at Day 30
Description: Phosphorylation (p): pSTAT3, pSTAT5 (Y694), and pS6 among Treg and non-Treg at day +30.
Time Frame: 30 days post HCT
Population: All participants.
Measure: Median (Full Range); unit: percentage in total CD4s
Arm/Group | GVHD Regimen
Number analyzed (Participants) | 20
percentage in total CD4s
  pSTAT3 | 34.1 [10.4 to 99.7]
  pSTAT5 | 97.1 [44 to 99.9]
  pS6 | 19.3 [13.8 to 41.1]

10. Secondary Outcome: STAT3, STAT5 (Y694), and S6 Phosphorylation Among Treg and Non-Treg at Day 90
Description: Phosphorylation (p): pSTAT3, pSTAT5 (Y694), and pS6 among Treg and non-Treg at day +90.
Time Frame: 90 days post HCT
Population: All participants.
Measure: Median (Full Range); unit: percentage in total CD4s
Arm/Group | GVHD Regimen
Number analyzed (Participants) | 20
percentage in total CD4s
  pSTAT3 | 20.2 [2.56 to 61.8]
  pSTAT5 | 78.6 [33.6 to 100]
  pS6 | 16.3 [0.91 to 26.6]

11. Other Pre Specified Outcome: Function of Blood Treg After Allogeneic HSCT
Description: Percent of Treg suppression at day +30. Investigators had also planned to test Treg function at day +90, if sufficient Tregs had been available for analysis.
Time Frame: 30 days post HCT
Population: All evaluable participants at day +30.
Measure: Median (Standard Deviation); unit: percentage of suppression
Arm/Group | GVHD Regimen
Number analyzed (Participants) | 3
percentage of suppression | 61.0 (11.15)

12. Other Pre Specified Outcome: Rate of Natural Killer Cell (NK) Reconstitution
Description: Investigators planned to monitor natural killer cell (NK) reconstitution. Standard immune deficiency flow cytometry panels (IDP) was to be drawn on days +90, +180, and +365 to evaluate NK reconstitution. Results of standard lab tests to be compared to compiled data at a later date
Time Frame: 365 days post HCT
Population: Lab test results to be compared to compiled data at a later date.
Arm/Group | GVHD Regimen
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years, 6 months
Arm/Group | GVHD Regimen
Serious Adverse Events (participants affected / at risk) | 11/20
Other Adverse Events (participants affected / at risk) | 4/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GVHD Regimen (N=20)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fever (General disorders) | 3 (3)
Pain (General disorders) | 1 (1)
Hepatobiliary disorders - Other, VOD (Hepatobiliary disorders) | 2 (2)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Infections and infestations - Other, pneumonia (Infections and infestations) | 1 (1)
Infections and infestations - Other, staphylococcus epidermis bacteremia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Cystitis non-infective (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, adenovirus cystitis (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, kidney stones (Renal and urinary disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GVHD Regimen (N=20)
Ileus (Gastrointestinal disorders) | 1 (1)
Hepatobiliary disorders - Other, portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Strategies to overcome interference from soluble IL-2 receptor and STAT3-mediated acute GVHD are needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes